CLINICAL TRIAL: NCT01007110
Title: The Effects of Docosahexaenoic Acid (DHA) on Fetal Cardiac Outcomes
Brief Title: Effects of Docosahexaenoic Acid (DHA) on Fetal Cardiac Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Kathleen Gustafson, Ph.D., Research Assistant Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 11625
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Pregnancy
Keywords: DHA
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosahexaenoic Acid (DHA) (Active Comparator): Docosahexaenoic Acid (DHA)
  Interventions: Dietary Supplement: DHA
- Placebo (Placebo Comparator): soy/corn oil placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: DHA — Docosahexaenoic Acid (DHA) from algal oil
  Other Names: Docosahexaenoic acid
  Arms: Docosahexaenoic Acid (DHA)
Other: Placebo — Placebo capsule
  Other Names: Algal oil
  Arms: Placebo

SUMMARY:
DHA, a type of fatty acid, is important in early development, both in terms of reproductive physiology of gestation and in postnatal behavioral and cognitive function. In adults, DHA has been shown to lower triglycerides and is important to cardiovascular health and autonomic control, lowering heart rate and blood pressure and increasing heart variability. Little is known about how fatty acids impact cardiac control in infants, children or the fetus. Our hypothesis is that maternal DHA supplementation (600 mg/day) will lower fetal HR and increase fetal HRV.

DETAILED DESCRIPTION:
We have observed that maternal DHA supplementation during pregnancy results in lower fetal heart rate (HR) and higher heart-rate variability (HRV). In another study, we found that infants on DHA supplemented formula have lower HR. Because DHA supplementation in infancy is associated with improved neurobehavioral outcomes and infants with lower HR and higher vagal control have been found to have improved developmental outcomes, the first aim is to conduct a randomized, placebo-controlled trial to determine whether maternal DHA supplementation during pregnancy results in lower HR and higher HRV in the fetal period. We will document other fetal neurobehaviors (body and breathing movements) as they are hallmarks of fetal well-being and influence HR and HRV.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females 16.0-35.99 years of age who are 12 to 20 weeks gestation at the time of enrollment (by dates or ultrasound)
* Agree to consume study capsules from enrollment until delivery
* BMI <40 at baseline or weight does not exceed 300 pounds
* No serious illnesses likely to confound study outcomes
* Available by phone

Exclusion Criteria:

* Less than 16 or greater than 35.99 years of age at enrollment
* BMI >40 at baseline
* Any serious illness likely to confound primary study outcomes
* Expecting multiple infants
* Diabetes (Type I, II or gestational) at baseline
* Elevated blood pressure due to any cause (systolic BP >= 140 mm Hg
* Gestational age at baseline < 12 weeks or > 20 weeks
* Unable to provide informed consent in English

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gustafson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Gustafson KM, Carlson SE, Colombo J, Yeh HW, Shaddy DJ, Li S, Kerling EH. Effects of docosahexaenoic acid supplementation during pregnancy on fetal heart rate and variability: a randomized clinical trial. Prostaglandins Leukot Essent Fatty Acids. 2013 May;88(5):331-8. doi: 10.1016/j.plefa.2013.01.009. Epub 2013 Feb 20. PMID 23433688
- [Derived] Christifano DN, Taylor MK, Carlson SE, Colombo J, Gustafson KM. Higher maternal weight is related to poorer fetal autonomic function. J Dev Orig Health Dis. 2021 Jun;12(3):354-356. doi: 10.1017/S2040174420000653. Epub 2020 Jul 14. PMID 32662379
- [Derived] Hoyer D, Schmidt A, Gustafson KM, Lobmaier SM, Lakhno I, van Leeuwen P, Cysarz D, Preisl H, Schneider U. Heart rate variability categories of fluctuation amplitude and complexity: diagnostic markers of fetal development and its disturbances. Physiol Meas. 2019 Jul 3;40(6):064002. doi: 10.1088/1361-6579/ab205f. PMID 31071684

RESULTS

PARTICIPANT FLOW:
Groups:
- Docosahexaenoic Acid (DHA): 600 mg Docosahexaenoic Acid (DHA)
Period: Allocation
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 32 | 35
Completed | 25 | 27
Not Completed | 7 | 8
Period: Follow-Up at 24 Weeks
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 25 | 27
Completed | 25 | 23
Not Completed | 0 | 4
Period: Follow-Up at 32 Weeks
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 25 | 23
Completed | 24 | 22
Not Completed | 1 | 1
Period: Follow-Up at 36 Weeks
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 24 | 22
Completed | 24 | 20
Not Completed | 0 | 2
Period: Neonatal Behavioral Assessment Scale (NB
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 24 | 20
Completed | 12 | 15
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Docosahexaenoic Acid (DHA) | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.8) | 25.5 (4.3) | 25.5 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 67
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67
Enrollment BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (7.0) | 26.8 (5.5) | 27.9 (6.21)
Education [Mean (Standard Deviation); unit: Years] | 13.9 (2.7) | 14.0 (3.1) | 14 (2.89)
Gestational Age (GA) [Mean (Standard Deviation); unit: Weeks] | 15.2 (3.7) | 13.6 (4.1) | 14.4 (3.88)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Mean fetal heart rate calculated from the magnetocardiogram recorded at 24, 32 and 36 weeks gestational age.
Time Frame: 24, 32 and 36 weeks gestational age
Population: Placebo: 19 subjects @ 24 wks GA, 25 subjects @ 32 wks GA, 24 subjects @ 36 wks GA
  DHA: 21 subjects @ 24 wks GA, 23 subjects @ 32 wks GA, 22 subjects @ 36 wks GA
Measure: Mean (Standard Deviation); unit: Beats per minute
Groups:
- Docosahexaenoic Acid (DHA): 600 mg/day docosahexaenoic acid (DHA)
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 25 | 23
Beats per minute
  Heart Rate 24 weeks Gestational Age | 146.0 (6.5) | 145.2 (6.8)
  Heart Rate 32 weeks Gestational Age | 142.5 (7.7) | 140.8 (7.6)
  Heart Rate 36 weeks Gestational Age | 145.0 (8.6) | 141.7 (9.3)

2. Secondary Outcome: Neonatal Behavioral Assessment Scale (NBAS) Scores
Description: The Neonatal Behavioral Assessment Scale (NBAS) measure 6 areas.
  For behavioral items a higher score corresponds to more desirable outcomes:
  1. Habituation: Sum of scores across 3 items, scored on a scale of 1-9. Range: 3-27.
  2. Orientation: Sum of scores across 7 items, scored on a scale of 1-9. Range: 7 - 63.
  3. Motor: Sum of scores across 5 items; 3 scored on a scale of 1-9, 1 scored on a scale of 1-6, and 1 scored on a scale of 1-5. Range: 5-38.
  4. Range of State: Sum of scores across 4 items; 2 scored on a scale of 1-6 and 2 scored on a scale of 1-5. Range: 4-22.
  5. Regulation of State: Sum of scores across 4 items, scored on a scale of 1-9. Range: is 4-36.
  6. Autonomic Stability: Sum of scores across 3 items; 1 scored on a scale of 1-9, 1 on a scale of 1-8, and 1 on a scale of 1-6. Range: 3-23.
  Reflexes: Sum across the 18 items, scored on a scale of 0-3. Range: 0 to 54. The supplementary items are each scored on a scale of 1-9 and do not combine to form a composite.
Time Frame: within 2 weeks of delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Docosahexaenoic Acid (DHA): 600 mg/day docosahexaenoic acid
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 12 | 15
units on a scale
  Habituation | 9.92 (9.28) | 8.47 (9.26)
  Orienting | 19.75 (15.45) | 23.40 (18.32)
  Motor | 23.08 (11.40) | 26.07 (18.13)
  State Organization | 13.50 (13.89) | 15.13 (8.02)
  State Regulation | 16.42 (20.02) | 16.93 (20.06)
  Autonomic | 14.83 (16.90) | 18.13 (14.48)
  Reflexes | 21.92 (14.45) | 22.60 (14.33)

3. Secondary Outcome: Maternal Red Blood Cell (RBC) Phospholipids at Delivery
Description: Maternal red blood cell phospholipid collected at delivery. These results were compared to baseline red blood cell phospholipid that was collected at study enrollment. A weighed standard fatty acid mixture (Supelco 37 component fatty acid methyl ester mix,Sigma Aldrich) was employed to correct final DHA weight percent of total fatty acids (wt%TFA).
Time Frame: Time of delivery, 36 weeks to term
Measure: Median (Inter-Quartile Range); unit: weight percent Total Fatty Acids
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 24 | 22
weight percent Total Fatty Acids | 4.99 [4.42 to 5.69] | 7.09 [5.39 to 10.3]

4. Secondary Outcome: Cord Blood Phospholipids DHA
Description: Newborn red blood cell phospholipids collected at birth.
Time Frame: Birth
Measure: Median (Inter-Quartile Range); unit: weight percent total fatty acids
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 24 | 22
weight percent total fatty acids | 6.18 [5.81 to 6.87] | 7.75 [6.01 to 9.03]

5. Secondary Outcome: Cardiac Conduction Time
Time Frame: Change from Baseline to 2 Months Post-natal
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 24 | 22
milliseconds | 38.98 (3.62) | 39.49 (2.798)

ADVERSE EVENTS:
Time Frame: Adverse Event Data were reviewed and reported by the Data Safety and Monitoring Board (DSMB) every 6 months for the 2 year duration of the study.
Description: Adverse events were categorized by body system affected by the study monitor (systematic assessment). Serious AEs were reported within 24 hours of their occurrence, AEs were reported every 3 months. The DSMB met every 6 months.
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes